CLINICAL TRIAL: NCT05775419
Title: A Prospective Randomized Controlled Clinical Study Comparing Curative Effect of Non-surgical Esophageal Squamous Cell Carcinoma With Radical Chemoradiotherapy and Radical Chemoradiotherapy Combined With Consolidation Chemotherapy
Brief Title: Comparison of Chemoradiotherapy and Chemoradiotherapy Combined With Consolidation Chemotherapy for ESCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GXL-003
Record Dates: First submitted 2022-09-07; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Esophageal Squamous Cell Carcinoma; Chemotherapy Effect; Side Effect of Drug
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Consolidation Chemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: radical chemoradiotherapy group; (Sham Comparator): Concurrent chemotherapy (2 courses): Lipusu (T) + Cisplatin (DDP) scheme: T 135mg/m2 ivgtt, d1, 3week*2cycles; DDP 75mg/m2 ivgtt, d2, 3week*2cycles; Radiotherapy scheme: intensity modulated radiotherapy PTV50-54Gy, PGTV 56-60Gy, conventional fractionation.
  Interventions: Combination Product: Concurrent chemotherapy (2 courses)
- Group B: radical chemoradiotherapy combined with consolidation chemotherapy group (Experimental): Consolidation chemotherapy (4 courses): After the concurrent chemoradiotherapy is over, after 2-3 weeks of rest, the patients in the consolidation chemotherapy group will be given 4 cycles of consolidation chemotherapy, and the chemotherapy regimen is the same as the concurrent chemotherapy regimen; Radiotherapy scheme: intensity modulated radiotherapy PTV50-54Gy, PGTV 56-60Gy, conventional fractionation.
  Interventions: Combination Product: Consolidation chemotherapy (4 courses)

INTERVENTIONS:
Combination Product: Consolidation chemotherapy (4 courses) — Consolidation chemotherapy (4 courses): After the concurrent chemoradiotherapy is over, after 2-3 weeks of rest, the patients in the consolidation chemotherapy group will be given 4 cycles of consolidation chemotherapy, and the chemotherapy regimen is the same as the concurrent chemotherapy regimen;
  Arms: Group B: radical chemoradiotherapy combined with consolidation chemotherapy group
Combination Product: Concurrent chemotherapy (2 courses) — Lipusu (T) + Cisplatin (DDP) program: T 135mg/m2 ivgtt, d1, 3week*2cycles; DDP 75mg/m2 ivgtt, d2, 3week*2cycles;
  Arms: Group A: radical chemoradiotherapy group;

SUMMARY:
This study is a phase III, multicenter, prospective randomized controlled clinical study comparing the efficacy of non-surgical esophageal squamous cell carcinoma with radical chemoradiotherapy and radical chemoradiotherapy combined with consolidation chemotherapy. The survival time and side effects of patients were observed and compared.

DETAILED DESCRIPTION:
Test grouping:

Group A: radical chemoradiotherapy group; Group B: radical chemoradiotherapy combined with consolidation chemotherapy group;

Specific chemotherapy regimens:

Concurrent chemotherapy (2 courses): Lipusu (T) + Cisplatin (DDP) scheme: T 135mg/m2 ivgtt, d1, 3week*2cycles; DDP 75mg/m2 ivgtt, d2, 3week*2cycles; Consolidation chemotherapy (4 courses): After the concurrent chemoradiotherapy is over, after 2-3 weeks of rest, the patients in the consolidation chemotherapy group will be given 4 cycles of consolidation chemotherapy, and the chemotherapy regimen is the same as the concurrent chemotherapy regimen; Radiotherapy scheme: intensity modulated radiotherapy PTV50-54Gy, PGTV 56-60Gy, conventional fractionation.

Primary efficacy endpoints: 3-year overall survival (OS), 5-year overall survival (OS) Secondary efficacy endpoints: 3-year progression-free survival (PFS), 5-year progression-free survival (PFS), objective response rate (ORR), disease control rate (DCR), toxic and side effects, and patient quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, not limited to male or female; at least able to take liquid diet;
2. Esophageal squamous cell carcinoma proved by histopathology;
3. Esophageal squamous cell carcinoma that is inoperable or refuses surgery,
4. According to the 2017 8th edition of AJCC esophageal cancer new staging criteria, the tumor is T2N0M0-TxNxM0 stage;
5. ECOG 0-1; life expectancy > 6 months;
6. No chemotherapy was used before selection;
7. No history of radiotherapy;
8. No surgical treatment;
9. No serious allergic history;
10. Hemoglobin 100 g/L, WBC3.5109/L, neutrophils 1.5109, platelets 100109/L; CR1.5 upper limit of normal, TB2.5 upper limit of normal, AST and ALT2.5 upper normal limit, AKP2.5 upper normal limit ; Be able to understand the research and have signed the informed consent;

Exclusion Criteria:

1. History of malignant tumors in other parts;
2. Duplicate carcinoma of the esophagus;
3. Pregnant or lactating patients;
4. Fertility but not using contraceptive measures;
5. Serious comorbidities: very high-risk hypertension, severe pulmonary function impairment, massive myocardial infarction, cardiac function ≥ grade II, mental history and severe diabetes;
6. During the active period of infectious diseases;
7. Participate in other clinical trials at present or within four weeks before enrollment;
8. Simultaneous treatment with other anti-cancer drugs (including anti-cancer traditional Chinese medicine);
9. After esophageal stent placement;
10. Cases with perforation tendency;
11. Have a history of organ transplantation.
12. Widespread metastases throughout the body, including lung, liver, bone, and intracranial metastases;
13. Known or suspected allergic to chemotherapy drugs; According to the judgment of the investigator, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1216 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
3-years overall survival (OS) | up to 3 years
  Overall survival was measured from the initiation of chemotherapy to the date of the last follow-up or death.
5-years overall survival (OS) | up to 5 years
  Overall survival was measured from the initiation of chemotherapy to the date of the last follow-up or death.

SECONDARY OUTCOMES:
3-year progression-free survival (PFS) | up to 3 years
  The PFS was calculated from the initiation of chemotherapy to the date of disease progression or death.
Objective response rate (ORR) Objective response rate (ORR) | through study completion, an average of 36 month
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission
5-year progression-free survival (PFS) | up to 5 years
  The PFS was calculated from the initiation of chemotherapy to the date of disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin GE, MM, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China